CLINICAL TRIAL: NCT05530837
Title: Characterization of Enterococcus Faecalis Endocarditis and Impact of Amoxicillin MIC Elevation on Patient Outcome
Acronym: ENDO_ENTERO
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO_ENTERO
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Infectious Endocarditis
MeSH Terms: conditions — Endocarditis, Subacute Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infective endocarditis is a complex infection that can be life-threatening. These infections also cause anatomical lesions that can be severe. Their management is complex and involves several disciplines: cardiology, bacteriologists, infectious diseases specialists, radiologists, nuclear medicine specialists, cardiac surgeons, neurologists, pharmacologists, etc. The incidence of Enterococcus faecalis endocarditis is increasing due to the aging of the population and the disappearance of rheumatic fever. The adequate management of these infections is complex and relies on the prolonged administration of high-dose antibiotics, classically the combination of amoxicillin and ceftriaxone. In the context of Streptococcal endocarditis, the impact of increasing the Minimum Inhibitory Concentration (MIC) of amoxicillin on patient mortality has been demonstrated but no study has yet examined the impact of increasing the MIC of amoxicillin on the outcome of patients treated for Enterococcus faecalis infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age with a diagnosis of Enterococcus faecalis infective endocarditis based on Duke criteria
* Patient hospitalized in one of the participating centers
* French-speaking patient

Exclusion Criteria:

* Patient with suspected infective endocarditis who does not meet Duke criteria
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of their data for this research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age with a diagnosis of Enterococcus faecalis infective endocarditis based on Duke criteria
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Describe the epidemiology and clinical presentations of patients with Enterococcus faecalis endocarditis | Month 1
  This outcome corresponds to the evaluation of factors associated with mortality in patients with Enterococcus faecalis endocarditis.

SECONDARY OUTCOMES:
Impact of increasing the minimum inhibitory concentrations of amoxicillin on the outcome of Enterococcus faecalis infective endocarditis | Month 1
  This outcome corresponds to the description of the epidemiology of Enterococcus faecalis endocarditis in France.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Hôpital de La Croix Rousse, Lyon
  - Groupe Hospitalier Paris Saint-Joseph, Paris

REFERENCES:
- [Background] Herrera-Hidalgo L, Lomas-Cabezas JM, Lopez-Cortes LE, Luque-Marquez R, Lopez-Cortes LF, Martinez-Marcos FJ, de la Torre-Lima J, Plata-Ciezar A, Hidalgo-Tenorio C, Garcia-Lopez MV, Vinuesa D, Gutierrez-Valencia A, Gil-Navarro MV, De Alarcon A. Ampicillin Plus Ceftriaxone Combined Therapy for Enterococcus faecalis Infective Endocarditis in OPAT. J Clin Med. 2021 Dec 21;11(1):7. doi: 10.3390/jcm11010007. PMID 35011748
- [Background] Marino A, Munafo A, Zagami A, Ceccarelli M, Campanella E, Cosentino F, Moscatt V, Cantarella G, Di Mauro R, Bernardini R, Nunnari G, Cacopardo B. Ampicillin plus ceftriaxone therapy against Enterococcus faecalis endocarditis: A case report, guidelines considerations, and literature review. IDCases. 2022 Mar 2;28:e01462. doi: 10.1016/j.idcr.2022.e01462. eCollection 2022. PMID 35265458
- [Background] Shah NH, Shutt KA, Doi Y. Ampicillin-Ceftriaxone vs Ampicillin-Gentamicin for Definitive Therapy of Enterococcus faecalis Infective Endocarditis: A Propensity Score-Matched, Retrospective Cohort Analysis. Open Forum Infect Dis. 2021 Mar 6;8(4):ofab102. doi: 10.1093/ofid/ofab102. eCollection 2021 Apr. PMID 34805443
- [Background] Pilmis B, Lourtet-Hascoet J, Barraud O, Piau C, Isnard C, Hery-Arnaud G, Amara M, Merens A, Farfour E, Thomas E, Jacquier H, Zahar JR, Bonnet E, Monnier AL; GMC Study Group. Be careful about MICs to amoxicillin for patients with Streptococci-related infective endocarditis. Int J Antimicrob Agents. 2019 Jun;53(6):850-854. doi: 10.1016/j.ijantimicag.2019.03.002. Epub 2019 Mar 7. PMID 30851401